CLINICAL TRIAL: NCT04691154
Title: A Phase 3, 2-Part, Open-Label Study to Evaluate the Safety and Tolerability of Liposomal Treprostinil Inhalation Suspension (L606) in Subjects With Pulmonary Arterial Hypertension or Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: A Phase 3 Study to Evaluate the Safety and Tolerability of L606 in Subjects With PAH or PH-ILD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI L606p3
Record Dates: First submitted 2020-12-21; First posted 2020-12-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension Due to Lung Diseases
Keywords: treprostinil; Pulmonary Arterial Hypertension; inhalation; Pulmonary Hypertension Due to Lung Diseases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Cohort A: Tyvaso stabilized PAH or PH-ILD patients Cohort B: Prostacyclin naive - PAH patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L606 (Experimental)
  Interventions: Combination Product: L606 inhalation suspension

INTERVENTIONS:
Combination Product: L606 inhalation suspension — L606 inhalation suspension

SUMMARY:
This Phase 3, 2-part, open-label, multicenter study aims to demonstrate the safety and tolerability of L606 in patients with PAH or PH-ILD. The study will determine the short-term and long-term safety and tolerability of L606 in this patient population.

DETAILED DESCRIPTION:
This Phase 3, 2-part, open-label, multicenter study aims to demonstrate the safety and tolerability of repeated doses of L606 in patients with PAH or PH-ILD.

Cohort A: Subjects with PAH or PH-ILD receiving prior stable doses of Tyvaso and willing to switch to L606.

Cohort B: Subjects with PAH (not initially on prostacyclin therapy) who are likely to receive clinical benefit from inhaled treprostinil based on the opinion of the investigator.

Cohort A subjects will sequentially participate in the Main Study Period (MSP) for 2 weeks and the Open Extension Period (OEP) for 46 weeks. Cohort B subjects will sequentially participate in the MSP for 12 weeks and the OEP for 36 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females ≥18 and ≤80 years of age.
2. Diagnosed with

   1. PAH belonging to at least 1 of the following subgroups of Group 1 pulmonary hypertension (PH) per European Society of Cardiology/European Respiratory Society Guidelines for the diagnosis and treatment of PH at least 1 year prior to screening. or
   2. PH-ILD Group 3 European Society of Cardiology/European Respiratory Society Guidelines for the diagnosis and treatment of PH. Subjects with Group 3 PH that is not related to underlying ILD are not eligible.
3. Subjects with PAH: Documentation of having PAH as confirmed by RHC meeting the following criteria:

   i. Mean PAP >20 mmHg. ii. Pulmonary arterial wedge pressure ≤15 mmHg. iii. Pulmonary vascular resistance >3 Wood units. Subjects with PH-ILD: Confirmation of the underlying ILD must be based on HRCT imaging with demonstration of diffuse parenchymal lung disease and documented by the Investigator or radiology report. Subjects may have any form of ILD or CPFE.
4. NYHA functional class II, III, or IV at the screening visit.
5. Can complete a screening 6MWD of ≥150 meters
6. For subjects with PAH: >65% of predicted and FEV1/FVC ratio >65% at screening. For subjects with PH-ILD: >40% of predicted and FEV1/FVC ratio >70% at screening.

Key Exclusion Criteria:

1. LVEF of ≤45% on a historical echocardiogram.
2. History of sleep apnea, or left-sided heart disease (including but not limited to aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, or coronary artery disease) per investigator's discretion.
3. Experienced an acute exacerbation of disease or hospitalization for any reason within 30 days of signing the ICF or prior to baseline.
4. Musculoskeletal disorder (eg, arthritis affecting the lower limbs, recent hip or knee joint replacement) or any disease that would likely be the primary limit to ambulation or subject is connected to a machine that is not portable enough to allow for a 6MWT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability assessed by incidence of treatment-emergent AEs/SAEs | 2 weeks
  (MSP for Cohort A): Proportion of patients with PAH or PH-ILD on a stable Tyvaso dose who would develop treatment-emergent AEs/SAEs after switching to L606 dosing for up to 2 weeks during MSP.
Safety/Tolerability assessed by incidence of treatment-emergent AEs/SAEs | 12 weeks
  (MSP for Cohort B): Proportion of patients with PAH (not initially on prostacyclin therapy) who would develop treatment-emergent AEs/SAEs during 12 weeks of the MSP with titration on twice daily L606.
Safety/Tolerability assessed by incidence of treatment-emergent AEs/SAEs (long-term) | 48 weeks
  (OEP for Cohorts A and B): Proportion of subjects with PAH or PH-ILD, choosing to continue twice daily L606 dosing for up to 48 weeks, who would develop treatment emergent AEs/SAEs up to 48 hours after the last dose.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Pulmonary Specialists, Scottsdale, Arizona
  - VA Greater Los Angeles Healthcare, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Summit Health Eastside Clinic, Bend, Oregon
  - Baylor Scott and White Research Institute, Temple, Texas